CLINICAL TRIAL: NCT01308307
Title: Is Non-cycloplegic Photorefraction Applicable for Screening Refractive Risk Factors of Amblyopia?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Zhale Rajavi, Ophthalmic Research center
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: 8821
Record Dates: First submitted 2011-03-03; First posted 2011-03-04 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2009-10

CONDITIONS: Amblyopia
Keywords: Non-cycloplegic photorefraction; cycloplegic refraction,; Amblyopia
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor

ARMS (1):
- one arm (Experimental)
  Interventions: Device: photorefraction

INTERVENTIONS:
Device: photorefraction — photorefraction is a name of device.

SUMMARY:
Purpose: : This study was performed to compare the accuracy of non-cycloplegic photorefraction with cycloplegic refraction in detection of refractive amblyopia risk factors and determine some corresponding beneficial cut points.

Method: In this diagnostic accuracy study, right eyes of 185 children (1 to 14 years) underwent first non-cycloplegic photorefraction (with PlusOptix SO4 photoscreener) and then cycloplegic refraction from October 2009 to August 2010. Based on the cycloplegic refraction results, hyperopia (≥+3.5D), myopia (≥-3D), astigmatism (≥1.5D), and anisometropia (≥1.5D) were set as criteria based on AAPOS guidelines. The difference in detection of refractive amblyopia risk factors between the two methods was the main outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* > 1 year old /with consent

Exclusion Criteria:

* mental retardation
* impaired fixation
* strabismus
* ptosis and any other organic ophthalmic disorder interfering with refraction

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 185 (Actual)
Dates: Start 2009-10; Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
refraction | 10 months
  cycloplegic auto refraction & Non-cycloplegic photorefraction

SECONDARY OUTCOMES:
hyperopia (≥+3.5D), myopia (≥-3D), astigmatism (≥1.5D), and anisometropia (≥1.5D) were set as criteria based on AAPOS guidelines. | 10 months
  cycloplegic auto refraction & Non-cycloplegic photorefraction

CONTACTS AND LOCATIONS:
Locations (1):
- Labbafinejad medical center, Tehran, Iran